CLINICAL TRIAL: NCT00766337
Title: A Phase 2, Randomized, Masked, Controlled Clinical Study to Assess the Safety and Efficacy of Lucentis® Plus Sirolimus Versus Lucentis® Plus Placebo in Patients With Sub-Foveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Phase 2 Study of an Ocular Sirolimus (Rapamycin) Formulation in Combination With Lucentis® in Patients With Age-Related Macular Degeneration
Acronym: EMERALD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMD-003
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2010-07

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: wet AMD
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Sirolimus; Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Group 1 (Experimental)
  Interventions: Drug: Sirolimus in combination with ranibizumab
- Dose Group 2 (Experimental)
  Interventions: Drug: Sirolimus in combination with ranibizumab
- Dose Group 3 (Placebo Comparator)
  Interventions: Drug: Placebo in combination with ranibizumab

INTERVENTIONS:
Drug: Sirolimus in combination with ranibizumab — Combination therapy of 440 micrograms sirolimus injected subconjunctivally and 500 micrograms ranibizumab injected intravitreally over a 60 day treatment period.
  Other Names: MS-R001; rapamycin; Lucentis
  Arms: Dose Group 1
Drug: Sirolimus in combination with ranibizumab — Combination therapy of 1320 micrograms sirolimus injected subconjunctivally and 500 micrograms ranibizumab injected intravitreally over a 60 day treatment period.
  Other Names: MS-R002; rapamycin; Lucentis
  Arms: Dose Group 2
Drug: Placebo in combination with ranibizumab — Combination therapy of placebo injected subconjunctivally and 500 micrograms ranibizumab injected intravitreally over a 60 day treatment period.
  Other Names: vehicle; Lucentis
  Arms: Dose Group 3

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an ocular sirolimus (rapamycin) formulation in combination with Lucentis in patients with sub-foveal choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sub-foveal choroidal neovascularization secondary to age-related macular degeneration within six months of initial study visit, and may have been treated with up to 3 Lucentis® (ranibizumab) or 3 Avastin® (bevacizumab) injections with the last injection administered at least 4 weeks prior to the initial study visit, or is treatment-naïve
* Visual acuity of 20/40 to 20/200 in the study eye

Exclusion Criteria:

* Any other ocular disease that could compromise vision in the study eye
* Presence of other causes of choroidal neovascularization other than secondary to age-related macular degeneration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity by ETDRS | 120 days

SECONDARY OUTCOMES:
Retinal thickness | 120 days
Safety across treatment groups | Through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Director — MacuSight, Inc.
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States